CLINICAL TRIAL: NCT06947668
Title: Immune Biomarker Study for Cisplatin-ineligible Patients Receiving Chemoradiotherapy With Docetaxel
Acronym: DoIT_Neck
Status: Not yet recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: DoIT_Neck
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Squamous Cell Carcinoma of Oropharynx; Squamous Cell Carcinoma of the Hypopharynx; Larynx Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumour tissue; stool sample; blood samples; saliva samples (mucosal swabs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: Patients with squamous cell carcinoma of the head and neck without distant metastases, for whom definitive or postoperative chemoradiation is indicated and who are unfit for cisplatin.

SUMMARY:
Analysis of tumor tissue (which is already available in pathology) and collection of saliva/stool and blood samples, which are obtained as part of a routine collection. These will be evaluated together with the patients' clinical data to identify possible predictors for treatment feasibility, survival, tumor control and potentially increased tumor immunogenicity by docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Patients with squamous cell carcinomas of the oropharynx, larynx and oral cavity for whom definitive or postoperative chemoradiation is indicated
* Patients who are cisplatin-unfit for chemotherapy, defined as:

  * ECOG 2
  * Organ dysfunction ≥ 2 according to National Cancer Institute Common Toxicity Criteria (NCI CTC) Version 4.0, such as hearing loss or tinnitus or neurological diseases
  * Calculated creatinine clearance of ≤50ml/min
  * Impaired organ function or comorbidities that preclude the use of cisplatin, e.g.: left ventricular ejection fraction < 50%, uncorrectable renal insufficiency with elevated creatinine despite creatinine clearance of 50ml/min due to increased body weight, uncontrolled hypertension
  * Poor nutritional status BMI < 16kg/m²
  * Concomitant use of nephrotoxic drugs that cannot be discontinued or converted due to other illnesses.
  * Willingness of patients to provide blood, saliva and stool samples and consent to the preservation of all samples for study purposes
  * Age ≥ 18 years
  * Sufficient cognitive abilities of the patients to understand the purpose of the study and to consent to it

Exclusion Criteria:

* Distant metastases at the time of diagnosis and simultaneous second cancers, i.e. at the time of study inclusion
* Malignancies in the last 5 years regardless of location (except basal cell carcinoma or cervical uteri)
* Carcinomas in which no sample collection is possible or likely without compromising the pathological assessment
* Persistent drug or medication abuse
* Patients who are unwilling or unable to comply with the protocol and receive treatment
* Patients who are unsuitable for participation in the study due to a language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with squamous cell carcinoma of the head and neck without distant metastases, for whom definitive or postoperative chemoradiation is indicated and who are unfit for cisplatin.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Determining the feasibility of simultaneous chemoradiotherapy with docetaxel in cisplatin-ineligible patients based on immunophenotype | 61 months (duration of entire trial)

SECONDARY OUTCOMES:
Correlation of immunophenotype with overall survival, locoregional control and side effects | 61 months (duration of entire trial)
Identification of immunological parameters associated with relevant treatment-related complications (e.g. infection, cytopenia) | 61 months (duration of entire trial)
Identification of patients who will benefit from immunotherapy. | 61 months (duration of entire trial)

OTHER OUTCOMES:
Identification of the point in time when immunotherapy should be used | 61 months (duration of entire trial)

CONTACTS AND LOCATIONS:
Overall Officials: Marlen Haderlein, MD, Principal Investigator — Universitätsklinikum Erlangen, Strahlenklinik
Locations (1):
- Universitätsklinikum Erlangen, Strahlenklinik, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No